CLINICAL TRIAL: NCT01079195
Title: Effectiveness and Tolerability of Tarka in the Treatment of Hypertensive Patients With High Risk of Developing Diabetes Mellitus, Not Controlled on Single-drug Therapy: A Multicountry, Multicenter, Post-marketing Observational Study in the Routine Clinical Use
Brief Title: Effectiveness and Tolerability of Tarka® in the Treatment of Hypertensive Patients With High Risk of Developing Diabetes Mellitus
Acronym: TARDIA
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Cornelia Preda MD/Medical Director Romania & Bulgaria, Abbott
Other Study IDs: P10-299
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Effectiveness and tolerability of Tarka; Hypertensive patients; Diabetes mellitus; Observational study
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Patient group with Hypertension: Single Patient group with Hypertension

SUMMARY:
The aim of this post-marketing observational study (PMOS) is to provide data on the effectiveness and tolerability of Tarka in patients with a high risk of developing diabetes mellitus, as prescribed by the physicians in a community setting and in accordance with the terms of the local marketing authorization. The following specific questions will be addressed:

* Effectiveness of Tarka in lowering the blood pressure in hypertensive patients being at high risk of developing diabetes, not controlled on single-drug therapy.
* Tolerability of Tarka as assessed by withdrawal rates.

DETAILED DESCRIPTION:
This is a non-interventional, observational, open-label, multicountry, multicenter post-marketing study in which Tarka is prescribed in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication. Patients with a high risk of developing diabetes mellitus treated by secondary care specialists (such as internal medicine specialists, nephrologists, endocrinologists, etc.), whose hypertension is not controlled on single-drug therapy will be included.

The assignment of the patient to the treatment with Tarka is not decided in advance by this protocol but falls within current practice. The prescription of Tarka is clearly separated from the decision to include the patient in this study. No additional procedures (other than standard of care) shall be applied to the patients.

Each patient will be treated at the physician's discretion. Dosing schedule should be in the accordance with the locally approved Summary of Product Characteristics (SmPC). Physicians will be provided with a study kit that includes a protocol, Tarka's locally approved SmPC, and case reports forms for each patient to be enrolled.

The patient's demographic data, height, weight and waist circumference will be reported in the Inclusion visit. The previous antihypertensive therapy should be noted (generic name of the drug and total daily dose). All other drugs the patient currently receives for cardiovascular disease treatment should be recorded as well.

The patient will then be followed via regular office visits as determined by the physician. As this study is observational in nature, patient follow-up is not interventional and is left to the judgment of each physician within the 6-month period, which defines the survey for each patient. For indicative purposes, follow-up of participant should enable 3 patient visits during this period. For these reasons, the most likely visits are defined as "Inclusion visit" at which treatment with Tarka is to be commenced, and then "Follow-up visit Month 3 " and "Follow-up visit Month 6", although dates will depend only on the decision of the physician. As a result, failure to meet these suggested dates will not constitute a breach of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either gender (more than 18 years of age), with established diagnosis of essential hypertension (systolic blood pressure/ diastolic blood pressure greater than 140/90 mmHg)
* Patients not controlled on single-drug therapy and decision was made to introduce Tarka
* Patients with a high risk of developing diabetes mellitus (defined according British Medical Society guidelines) with at least one of the following symptoms:

  * Positive family history of diabetes or
  * Obesity defined by a Body Mass Index (BMI) greater than 30 kg/m^2 or a waist circumference greater than 102 cm (males) or greater than 88 cm (females) or
  * Impaired fasting plasma glucose (FPG) levels of 6.1 to 7.0 mmol/l (100-126 mg/dl)

Exclusion Criteria:

* Patients with known or established Type 2 diabetes mellitus
* The use of Tarka is contraindicated in the following patients:

  * Hypersensitive to the active substances or to any of the inactive ingredients
  * With cardiogenic shock
  * With second and third degree atrioventricular block - except in patients with a functioning artificial pacemaker
  * With sick sinus syndrome - except in patients with a functioning artificial pacemaker
  * With atrial fibrillation/flutter and concomitant Wolff-Parkinson-White syndrome
  * With existing history of angioedema associated with administration of an angiotensin-converting enzyme (ACE) inhibitor
  * With severe renal or severe liver impairment
  * In pregnant women (women of childbearing potential who are unwilling to use contraception should not be included)
  * Lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a high risk of developing diabetes mellitus treated by secondary care specialists (such as internal medicine specialists, nephrologists, endocrinologists, etc.), whose hypertension is not controlled on single-drug therapy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 15436 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Preda, MD, Study Director — Abbott International
Locations (898):
- Bulgaria (15):
  - Site Reference ID/Investigator# 29197, Haskovo
  - Site Reference ID/Investigator# 29685, Pleven
  - Site Reference ID/Investigator# 29682, Plovdiv
  - Site Reference ID/Investigator# 29686, Plovdiv
  - Site Reference ID/Investigator# 29097, Sofia
  - Site Reference ID/Investigator# 28954, Sofia
  - Site Reference ID/Investigator# 29681, Sofia
  - Site Reference ID/Investigator# 29683, Sofia
  - Site Reference ID/Investigator# 29079, Sofia
  - Site Reference ID/Investigator# 29651, Sofia
  - Site Reference ID/Investigator# 29484, Stara Zagora
  - Site Reference ID/Investigator# 29485, Stara Zagora
  - Site Reference ID/Investigator# 29480, Varna
  - Site Reference ID/Investigator# 7568, Varna
  - Site Reference ID/Investigator# 29196, Veliko Tarnovo
- Czechia (304):
  - Site Reference ID/Investigator# 28887, Adamov
  - Site Reference ID/Investigator# 28660, Aš
  - Site Reference ID/Investigator# 28705, Aš
  - Site Reference ID/Investigator# 28726, Bílina
  - Site Reference ID/Investigator# 29013, Bílina
  - Site Reference ID/Investigator# 29146, Bílina
  - Site Reference ID/Investigator# 29070, Bohumín
  - Site Reference ID/Investigator# 28891, Bolatice
  - Site Reference ID/Investigator# 28803, Boršov nad Vltavou
  - Site Reference ID/Investigator# 29047, Boskovice
  - Site Reference ID/Investigator# 29108, Brandýsek
  - Site Reference ID/Investigator# 28843, Brasy-Stupno
  - Site Reference ID/Investigator# 28578, Brno
  - Site Reference ID/Investigator# 28737, Brno
  - Site Reference ID/Investigator# 29043, Brno
  - Site Reference ID/Investigator# 28706, Brno
  - Site Reference ID/Investigator# 28973, Brno
  - Site Reference ID/Investigator# 29173, Brno
  - Site Reference ID/Investigator# 29175, Brno
  - Site Reference ID/Investigator# 28908, Brno
  - Site Reference ID/Investigator# 29123, Brno
  - Site Reference ID/Investigator# 28759, Brno
  - Site Reference ID/Investigator# 28914, Brno
  - Site Reference ID/Investigator# 29117, Brno
  - Site Reference ID/Investigator# 29124, Brno
  - Site Reference ID/Investigator# 29134, Brno
  - Site Reference ID/Investigator# 28971, Brno
  - Site Reference ID/Investigator# 28972, Brno
  - Site Reference ID/Investigator# 29036, Brno
  - Site Reference ID/Investigator# 29044, Brno
  - Site Reference ID/Investigator# 29693, Broumov
  - Site Reference ID/Investigator# 29694, Broumov
  - Site Reference ID/Investigator# 28646, Břeclav
  - Site Reference ID/Investigator# 28874, Buštěhrad
  - Site Reference ID/Investigator# 28684, Cheb
  - Site Reference ID/Investigator# 28751, Cheb
  - Site Reference ID/Investigator# 28847, Cheb
  - Site Reference ID/Investigator# 29132, Cheb
  - Site Reference ID/Investigator# 29142, Cheb
  - Site Reference ID/Investigator# 28669, Chomutov
  - Site Reference ID/Investigator# 28732, Chrudim
  - Site Reference ID/Investigator# 28792, Chrudim
  - Site Reference ID/Investigator# 29017, Chrudim
  - Site Reference ID/Investigator# 29136, Čelákovice
  - Site Reference ID/Investigator# 28814, Černošín
  - Site Reference ID/Investigator# 29069, Červená Voda
  - Site Reference ID/Investigator# 28900, Česká Třebová
  - Site Reference ID/Investigator# 28634, České Budějovice
  - Site Reference ID/Investigator# 28651, České Budějovice
  - Site Reference ID/Investigator# 28798, České Budějovice
  - Site Reference ID/Investigator# 28877, České Budějovice
  - Site Reference ID/Investigator# 29118, Český Těšín
  - Site Reference ID/Investigator# 28854, Čistá
  - Site Reference ID/Investigator# 28696, Děčín
  - Site Reference ID/Investigator# 28748, Děčín
  - Site Reference ID/Investigator# 28852, Děčín
  - Site Reference ID/Investigator# 28936, Dolní Kalná
  - Site Reference ID/Investigator# 28786, Domažlice
  - Site Reference ID/Investigator# 28821, Domažlice
  - Site Reference ID/Investigator# 29021, Domažlice
  - Site Reference ID/Investigator# 28855, Duchcov
  - Site Reference ID/Investigator# 29139, Frenštát pod Radhoštěm
  - Site Reference ID/Investigator# 29158, Frýdek-Místek
  - Site Reference ID/Investigator# 28682, Frýdlant nad Ostravicí
  - Site Reference ID/Investigator# 28817, Havířov
  - Site Reference ID/Investigator# 28657, Havlíčkův Brod
  - Site Reference ID/Investigator# 28733, Havlíčkův Brod
  - Site Reference ID/Investigator# 28858, Hněvotín
  - Site Reference ID/Investigator# 28904, Horšovský Týn
  - Site Reference ID/Investigator# 28894, Hostinné
  - Site Reference ID/Investigator# 28665, Hranice
  - Site Reference ID/Investigator# 28700, Hranice
  - Site Reference ID/Investigator# 28809, Hranice
  - Site Reference ID/Investigator# 28933, Hranice
  - Site Reference ID/Investigator# 29155, Jablonec nad Nisou
  - Site Reference ID/Investigator# 28861, Jablonec nad Nisou
  - Site Reference ID/Investigator# 28630, Javorník
  - Site Reference ID/Investigator# 28648, Jihlava
  - Site Reference ID/Investigator# 28756, Jihlava
  - Site Reference ID/Investigator# 28836, Jihlava
  - Site Reference ID/Investigator# 28643, Jindřichův Hradec
  - Site Reference ID/Investigator# 28788, Jindřichův Hradec
  - Site Reference ID/Investigator# 28678, Karlovy Vary
  - Site Reference ID/Investigator# 28741, Karlovy Vary
  - Site Reference ID/Investigator# 28893, Karlovy Vary
  - Site Reference ID/Investigator# 28652, Kdyně
  - Site Reference ID/Investigator# 28796, Kladeruby
  - Site Reference ID/Investigator# 28645, Kladno
  - Site Reference ID/Investigator# 28916, Kladno
  - Site Reference ID/Investigator# 28647, Klatovy
  - Site Reference ID/Investigator# 28659, Klatovy
  - Site Reference ID/Investigator# 28773, Kolín
  - Site Reference ID/Investigator# 29156, Kolín
  - Site Reference ID/Investigator# 29393, Krnov
  - Site Reference ID/Investigator# 28872, Kroměříž
  - Site Reference ID/Investigator# 28760, Kunovice
  - Site Reference ID/Investigator# 28857, Kutná Hora
  - Site Reference ID/Investigator# 28886, Kutná Hora
  - Site Reference ID/Investigator# 28655, Lázně Bělohrad
  - Site Reference ID/Investigator# 28898, Lednice
  - Site Reference ID/Investigator# 29019, Liberec
  - Site Reference ID/Investigator# 29141, Libice nad Cidlinou
  - Site Reference ID/Investigator# 28723, Libušín
  - Site Reference ID/Investigator# 29153, Lipník nad Bečvou
  - Czech Republic Site Reference ID/Investigator# 28769, Litoměřice
  - Site Reference ID/Investigator# 28815, Litoměřice
  - Site Reference ID/Investigator# 29116, Litomyšl
  - Site Reference ID/Investigator# 29020, Lovosice
  - Site Reference ID/Investigator# 28650, Mariánské Lázně
  - Site Reference ID/Investigator# 28878, Mělník
  - Site Reference ID/Investigator# 29149, Městec Králové
  - Site Reference ID/Investigator# 28820, Mikulov
  - Site Reference ID/Investigator# 28824, Mimoň
  - Site Reference ID/Investigator# 28853, Mnichovo Hradiště
  - Site Reference ID/Investigator# 28867, Mohelnice
  - Site Reference ID/Investigator# 29361, Mohelnice
  - Site Reference ID/Investigator# 28662, Náchod
  - Site Reference ID/Investigator# 29128, Neratovice
  - Site Reference ID/Investigator# 29057, Nové Město nad Metují
  - Site Reference ID/Investigator# 28888, Nový Bor
  - Site Reference ID/Investigator# 28875, Nový Bydžov
  - Site Reference ID/Investigator# 28740, Nymburk
  - Site Reference ID/Investigator# 29695, Olomouc
  - Site Reference ID/Investigator# 29689, Olomouc
  - Site Reference ID/Investigator# 29692, Olomouc
  - Site Reference ID/Investigator# 29121, Opava
  - Site Reference ID/Investigator# 29688, Opočno
  - Site Reference ID/Investigator# 29071, Orlová
  - Site Reference ID/Investigator# 29014, Ostrava
  - Site Reference ID/Investigator# 28708, Ostrava
  - Site Reference ID/Investigator# 28746, Ostrava
  - Site Reference ID/Investigator# 28755, Ostrava
  - Site Reference ID/Investigator# 28863, Ostrava
  - Site Reference ID/Investigator# 29046, Ostrava
  - Site Reference ID/Investigator# 29691, Ostrava
  - Site Reference ID/Investigator# 28807, Ostrava
  - Site Reference ID/Investigator# 28868, Ostrava
  - Site Reference ID/Investigator# 29113, Ostrava
  - Site Reference ID/Investigator# 29690, Ostrava
  - Site Reference ID/Investigator# 28679, Ostrava
  - Site Reference ID/Investigator# 28664, Ostrava
  - Site Reference ID/Investigator# 28681, Ostrava
  - Site Reference ID/Investigator# 29152, Ostrava
  - Site Reference ID/Investigator# 28816, Ostrava
  - Site Reference ID/Investigator# 28711, Ostrava
  - Site Reference ID/Investigator# 28787, Ostrava
  - Site Reference ID/Investigator# 28905, Ostrava-Hostalkovice
  - Site Reference ID/Investigator# 28780, Ostrava-Krasne Pole
  - Site Reference ID/Investigator# 28663, Ostrava-Poruba
  - Site Reference ID/Investigator# 28902, Ostrov
  - Site Reference ID/Investigator# 28728, Otrokovice
  - Site Reference ID/Investigator# 28661, Pardubice
  - Site Reference ID/Investigator# 28668, Pardubice
  - Site Reference ID/Investigator# 28735, Pardubice
  - Site Reference ID/Investigator# 28742, Pardubice
  - Site Reference ID/Investigator# 28770, Pardubice
  - Site Reference ID/Investigator# 28776, Pardubice
  - Site Reference ID/Investigator# 28789, Pardubice
  - Site Reference ID/Investigator# 28845, Pardubice
  - Site Reference ID/Investigator# 28873, Pardubice
  - Site Reference ID/Investigator# 28964, Pardubice
  - Site Reference ID/Investigator# 29120, Pardubice
  - Site Reference ID/Investigator# 28777, Paseka
  - Site Reference ID/Investigator# 28615, Pelhřimov
  - Site Reference ID/Investigator# 28675, Pelhřimov
  - Site Reference ID/Investigator# 28670, Pilsen
  - Site Reference ID/Investigator# 28931, Pilsen
  - Site Reference ID/Investigator# 28685, Pilsen
  - Site Reference ID/Investigator# 29145, Pilsen
  - Site Reference ID/Investigator# 28683, Pilsen
  - Site Reference ID/Investigator# 28680, Pilsen
  - Site Reference ID/Investigator# 28827, Pilsen
  - Site Reference ID/Investigator# 28752, Pilsen
  - Site Reference ID/Investigator# 28785, Pilsen
  - Site Reference ID/Investigator# 28844, Písek
  - Site Reference ID/Investigator# 29143, Písek
  - Site Reference ID/Investigator# 29115, Planá nad Lužnicí
  - Site Reference ID/Investigator# 28676, Polička
  - Site Reference ID/Investigator# 28658, Postoloprty
  - Site Reference ID/Investigator# 28833, Prachatice
  - Site Reference ID/Investigator# 28703, Prague
  - Site Reference ID/Investigator# 28801, Prague
  - Site Reference ID/Investigator# 29060, Prague
  - Site Reference ID/Investigator# 28656, Prague
  - Site Reference ID/Investigator# 28623, Prague
  - Site Reference ID/Investigator# 28633, Prague
  - Site Reference ID/Investigator# 28698, Prague
  - Site Reference ID/Investigator# 28842, Prague
  - Site Reference ID/Investigator# 28802, Prague
  - Site Reference ID/Investigator# 29696, Prague
  - Site Reference ID/Investigator# 28790, Prague
  - Site Reference ID/Investigator# 28876, Prague
  - Site Reference ID/Investigator# 28687, Prague
  - Site Reference ID/Investigator# 28794, Prague
  - Site Reference ID/Investigator# 28631, Prague
  - Site Reference ID/Investigator# 28635, Prague
  - Site Reference ID/Investigator# 28797, Prague
  - Site Reference ID/Investigator# 28926, Prague
  - Site Reference ID/Investigator# 28767, Prague
  - Site Reference ID/Investigator# 28826, Prague
  - Site Reference ID/Investigator# 28831, Prague
  - Site Reference ID/Investigator# 28864, Prague
  - Site Reference ID/Investigator# 29376, Prague
  - Site Reference ID/Investigator# 29377, Prague
  - Site Reference ID/Investigator# 28617, Prague
  - Site Reference ID/Investigator# 28627, Prague
  - Site Reference ID/Investigator# 28649, Prague
  - Site Reference ID/Investigator# 28813, Prague
  - Site Reference ID/Investigator# 28840, Prague
  - Site Reference ID/Investigator# 29127, Prague
  - Site Reference ID/Investigator# 29396, Prague
  - Site Reference ID/Investigator# 29687, Prague
  - Site Reference ID/Investigator# 28913, Prague
  - Site Reference ID/Investigator# 28765, Prague
  - Site Reference ID/Investigator# 28928, Prague
  - Site Reference ID/Investigator# 28673, Prague
  - Site Reference ID/Investigator# 28795, Prague
  - Site Reference ID/Investigator# 28882, Prague
  - Site Reference ID/Investigator# 28911, Prague
  - Site Reference ID/Investigator# 28935, Prague
  - Site Reference ID/Investigator# 29150, Prague
  - Site Reference ID/Investigator# 28653, Prague
  - Site Reference ID/Investigator# 28823, Prague
  - Site Reference ID/Investigator# 28724, Prague
  - Site Reference ID/Investigator# 29131, Prague
  - Site Reference ID/Investigator# 28774, Prague
  - Site Reference ID/Investigator# 28692, Prague
  - Site Reference ID/Investigator# 29022, Pribram V-Zdabor
  - Site Reference ID/Investigator# 29111, Prostějov
  - Site Reference ID/Investigator# 29418, Prostějov
  - Site Reference ID/Investigator# 29420, Prostějov
  - Site Reference ID/Investigator# 28701, Přelouč
  - Site Reference ID/Investigator# 28822, Přelouč
  - Site Reference ID/Investigator# 28719, Přerov
  - Site Reference ID/Investigator# 28750, Přimda
  - Site Reference ID/Investigator# 28783, Příbram
  - Site Reference ID/Investigator# 28707, Rakovník
  - Site Reference ID/Investigator# 28768, Rakovník
  - Site Reference ID/Investigator# 29024, Rakovník
  - Site Reference ID/Investigator# 28714, Rosice
  - Site Reference ID/Investigator# 7575, Rosice
  - Site Reference ID/Investigator# 28772, Rožnov pod Radhoštěm
  - Site Reference ID/Investigator# 29137, Rožnov pod Radhoštěm
  - Site Reference ID/Investigator# 28674, Rybitví
  - Site Reference ID/Investigator# 28846, Řevnice
  - Site Reference ID/Investigator# 29300, Řevnice
  - Site Reference ID/Investigator# 28848, Sezimovo Ústí
  - Site Reference ID/Investigator# 28866, Sezimovo Ústí
  - Site Reference ID/Investigator# 29122, Slaný
  - Site Reference ID/Investigator# 28712, Slavičín
  - Site Reference ID/Investigator# 28628, Sokolov
  - Site Reference ID/Investigator# 28860, Sokolov
  - Site Reference ID/Investigator# 29067, Svitavy
  - Site Reference ID/Investigator# 28791, Štěpánkovice
  - Site Reference ID/Investigator# 28890, Šumperk
  - Site Reference ID/Investigator# 29066, Šumperk
  - Site Reference ID/Investigator# 28677, Tábor
  - Site Reference ID/Investigator# 28710, Tábor
  - Site Reference ID/Investigator# 28672, Telč
  - Site Reference ID/Investigator# 28704, Teplice
  - Site Reference ID/Investigator# 28811, Teplice
  - Site Reference ID/Investigator# 28862, Teplice
  - Site Reference ID/Investigator# 28758, Trhové Sviny
  - Site Reference ID/Investigator# 29157, Trinec-Kanada
  - Site Reference ID/Investigator# 28899, Trutnov
  - Site Reference ID/Investigator# 29110, Trutnov
  - Site Reference ID/Investigator# 28912, Třebíč
  - Site Reference ID/Investigator# 29126, Třebíč
  - Site Reference ID/Investigator# 28616, Třebíč
  - Site Reference ID/Investigator# 28739, Turnov
  - Site Reference ID/Investigator# 28747, Turnov
  - Site Reference ID/Investigator# 28925, Týn nad Vltavou
  - Site Reference ID/Investigator# 28927, Týn nad Vltavou
  - Site Reference ID/Investigator# 29151, Uherské Hradiště
  - Site Reference ID/Investigator# 28636, Újezd u Brna
  - Site Reference ID/Investigator# 29135, Újezd u Brna
  - Site Reference ID/Investigator# 28699, Ústí nad Labem
  - Site Reference ID/Investigator# 28869, Ústí nad Labem
  - Site Reference ID/Investigator# 29114, Ústí nad Orlicí
  - Site Reference ID/Investigator# 28709, Valašské Klobouky
  - Site Reference ID/Investigator# 28865, Valašské Meziříčí
  - Site Reference ID/Investigator# 28654, Valašské Meziříčí
  - Site Reference ID/Investigator# 29112, Valašské Meziříčí
  - Site Reference ID/Investigator# 29144, Valašské Meziříčí
  - Site Reference ID/Investigator# 28818, Vamberk
  - Site Reference ID/Investigator# 28895, Velké Hamry
  - Site Reference ID/Investigator# 29390, Vintířov
  - Site Reference ID/Investigator# 28713, Višňova
  - Site Reference ID/Investigator# 28624, Vlašim
  - Site Reference ID/Investigator# 29025, Vodňany
  - Site Reference ID/Investigator# 29018, Votice-Otradovice
  - Site Reference ID/Investigator# 29148, Vratimov
  - Site Reference ID/Investigator# 28666, Vsetín
  - Site Reference ID/Investigator# 28856, Vsetín
  - Site Reference ID/Investigator# 29109, Vsetín
  - Site Reference ID/Investigator# 29049, Vysoké Mýto
  - Site Reference ID/Investigator# 28697, Zahrádky
  - Site Reference ID/Investigator# 28837, Zábřeh
  - Site Reference ID/Investigator# 28781, Znojmo
  - Site Reference ID/Investigator# 28924, Znojmo
  - Site Reference ID/Investigator# 28804, Znojmo
  - Site Reference ID/Investigator# 28962, Žamberk
  - Site Reference ID/Investigator# 28906, Žďár
  - Site Reference ID/Investigator# 29048, Žirovnice
- Romania (42):
  - Site Reference ID/Investigator# 28575, Alba Iulia
  - Site Reference ID/Investigator# 28581, Bacau
  - Site Reference ID/Investigator# 28580, Bacau
  - Site Reference ID/Investigator# 29749, Baia Mare
  - Site Reference ID/Investigator# 29077, Brasov
  - Site Reference ID/Investigator# 32095, Bucharest
  - Site Reference ID/Investigator# 32096, Bucharest
  - Site Reference ID/Investigator# 28577, Bucharest
  - Site Reference ID/Investigator# 28605, Bucharest
  - Site Reference ID/Investigator# 29072, Bucharest
  - Site Reference ID/Investigator# 29073, Bucharest
  - Site Reference ID/Investigator# 28982, Bucharest
  - Site Reference ID/Investigator# 28955, Bucharest
  - Site Reference ID/Investigator# 28583, Buzău
  - Site Reference ID/Investigator# 32109, Cluj-Napoca
  - Site Reference ID/Investigator# 32110, Cluj-Napoca
  - Site Reference ID/Investigator# 32111, Cluj-Napoca
  - Site Reference ID/Investigator# 29099, Constanța
  - Site Reference ID/Investigator# 28579, Constanța
  - Site Reference ID/Investigator# 28584, Constanța
  - Site Reference ID/Investigator# 28992, Covasna
  - Site Reference ID/Investigator# 28613, Giurgiu
  - Site Reference ID/Investigator# 29074, Iași
  - Site Reference ID/Investigator# 28602, Iași
  - Site Reference ID/Investigator# 28967, Iași
  - Site Reference ID/Investigator# 28961, Odorheiu Secuiesc
  - Site Reference ID/Investigator# 28963, Oradea
  - Site Reference ID/Investigator# 29752, Oradea
  - Site Reference ID/Investigator# 28995, Piteşti
  - Site Reference ID/Investigator# 29628, Piteşti
  - Site Reference ID/Investigator# 29629, Piteşti
  - Site Reference ID/Investigator# 29031, Ploieşti
  - Site Reference ID/Investigator# 29191, Reşiţa
  - Site Reference ID/Investigator# 6369, Sibiu
  - Site Reference ID/Investigator# 29006, Suceava
  - Site Reference ID/Investigator# 29088, Târgovişte
  - Site Reference ID/Investigator# 29089, Târgu Mureş
  - Site Reference ID/Investigator# 29330, Târgu Mureş
  - Site Reference ID/Investigator# 29331, Târgu Mureş
  - Site Reference ID/Investigator# 29032, Tg. Mures
  - Site Reference ID/Investigator# 29087, Timișoara
  - Site Reference ID/Investigator# 29086, Timișoara
- Russia (190):
  - Site Reference ID/Investigator# 28596, Chelyabinsk
  - Site Reference ID/Investigator# 28986, Chelyabinsk
  - Site Reference ID/Investigator# 29248, Chelyabinsk
  - Site Reference ID/Investigator# 29332, Chelyabinsk
  - Site Reference ID/Investigator# 29546, Chelyabinsk
  - Site Reference ID/Investigator# 29547, Chelyabinsk
  - Site Reference ID/Investigator# 29491, Dmitrov
  - Site Reference ID/Investigator# 29492, Dmitrov
  - Site Reference ID/Investigator# 29496, Ivanteyevka
  - Site Reference ID/Investigator# 29221, Kazan'
  - Site Reference ID/Investigator# 29256, Kazan'
  - Site Reference ID/Investigator# 29423, Kazan'
  - Site Reference ID/Investigator# 29427, Kazan'
  - Site Reference ID/Investigator# 29562, Kazan'
  - Site Reference ID/Investigator# 29649, Kazan'
  - Site Reference ID/Investigator# 29650, Kazan'
  - Site Reference ID/Investigator# 28597, Kemerovo
  - Site Reference ID/Investigator# 29162, Kemerovo
  - Site Reference ID/Investigator# 29189, Kemerovo
  - Site Reference ID/Investigator# 29326, Kemerovo
  - Site Reference ID/Investigator# 29343, Kemerovo
  - Site Reference ID/Investigator# 29429, Kemerovo
  - Site Reference ID/Investigator# 29431, Kemerovo
  - Site Reference ID/Investigator# 29498, Khimki
  - Site Reference ID/Investigator# 28598, Korolyov
  - Site Reference ID/Investigator# 29499, Krasnodar
  - Site Reference ID/Investigator# 29500, Krasnodar
  - Site Reference ID/Investigator# 29501, Krasnodar
  - Site Reference ID/Investigator# 29502, Krasnodar
  - Site Reference ID/Investigator# 29503, Krasnodar
  - Site Reference ID/Investigator# 29504, Krasnodar
  - Site Reference ID/Investigator# 29527, Krasnogorsk
  - Site Reference ID/Investigator# 29530, Krasnogorsk
  - Site Reference ID/Investigator# 28979, Krasnoyarsk
  - Site Reference ID/Investigator# 28981, Krasnoyarsk
  - Site Reference ID/Investigator# 29174, Krasnoyarsk
  - Site Reference ID/Investigator# 29209, Krasnoyarsk
  - Site Reference ID/Investigator# 29444, Krasnoyarsk
  - Site Reference ID/Investigator# 29446, Krasnoyarsk
  - Site Reference ID/Investigator# 29448, Krasnoyarsk
  - Site Reference ID/Investigator# 29449, Krasnoyarsk
  - Site Reference ID/Investigator# 29451, Krasnoyarsk
  - Site Reference ID/Investigator# 29169, Lipetsk
  - Site Reference ID/Investigator# 29231, Lipetsk
  - Site Reference ID/Investigator# 28593, Moscow
  - Site Reference ID/Investigator# 28940, Moscow
  - Site Reference ID/Investigator# 28941, Moscow
  - Site Reference ID/Investigator# 28949, Moscow
  - Site Reference ID/Investigator# 28980, Moscow
  - Site Reference ID/Investigator# 29078, Moscow
  - Site Reference ID/Investigator# 29181, Moscow
  - Site Reference ID/Investigator# 29185, Moscow
  - Site Reference ID/Investigator# 29194, Moscow
  - Site Reference ID/Investigator# 29205, Moscow
  - Site Reference ID/Investigator# 29216, Moscow
  - Site Reference ID/Investigator# 29220, Moscow
  - Site Reference ID/Investigator# 29223, Moscow
  - Site Reference ID/Investigator# 29227, Moscow
  - Site Reference ID/Investigator# 29237, Moscow
  - Site Reference ID/Investigator# 29561, Moscow
  - Site Reference ID/Investigator# 29602, Moscow
  - Site Reference ID/Investigator# 29603, Moscow
  - Site Reference ID/Investigator# 29621, Moscow
  - Site Reference ID/Investigator# 29625, Mytischi
  - Site Reference ID/Investigator# 29532, N.Novgorod
  - Site Reference ID/Investigator# 29533, N.Novgorod
  - Site Reference ID/Investigator# 29534, N.Novgorod
  - Site Reference ID/Investigator# 29535, N.Novgorod
  - Site Reference ID/Investigator# 29634, N.Novgorod
  - Site Reference ID/Investigator# 29182, Novokuybyshevsk
  - Site Reference ID/Investigator# 29226, Novosibirsk
  - Site Reference ID/Investigator# 29536, Novosibirsk
  - Site Reference ID/Investigator# 29568, Novosibirsk
  - Site Reference ID/Investigator# 29619, Novosibirsk
  - Site Reference ID/Investigator# 29627, Novosibirsk
  - Site Reference ID/Investigator# 29647, Novosibirsk
  - Site Reference ID/Investigator# 29648, Novosibirsk
  - Site Reference ID/Investigator# 28592, Omsk
  - Site Reference ID/Investigator# 28976, Omsk
  - Site Reference ID/Investigator# 28977, Omsk
  - Site Reference ID/Investigator# 29335, Omsk
  - Site Reference ID/Investigator# 29337, Omsk
  - Site Reference ID/Investigator# 29338, Omsk
  - Site Reference ID/Investigator# 29339, Omsk
  - Site Reference ID/Investigator# 29537, Omsk
  - Site Reference ID/Investigator# 29622, Omsk
  - Site Reference ID/Investigator# 29511, Rostov-on-Don
  - Site Reference ID/Investigator# 29512, Rostov-on-Don
  - Site Reference ID/Investigator# 29513, Rostov-on-Don
  - Site Reference ID/Investigator# 29514, Rostov-on-Don
  - Site Reference ID/Investigator# 29515, Rostov-on-Don
  - Site Reference ID/Investigator# 29516, Rostov-on-Don
  - Site Reference ID/Investigator# 28594, Saint Petersburg
  - Site Reference ID/Investigator# 28603, Saint Petersburg
  - Site Reference ID/Investigator# 28942, Saint Petersburg
  - Site Reference ID/Investigator# 29178, Saint Petersburg
  - Site Reference ID/Investigator# 29200, Saint Petersburg
  - Site Reference ID/Investigator# 29210, Saint Petersburg
  - Site Reference ID/Investigator# 29213, Saint Petersburg
  - Site Reference ID/Investigator# 29217, Saint Petersburg
  - Site Reference ID/Investigator# 29246, Saint Petersburg
  - Site Reference ID/Investigator# 29341, Saint Petersburg
  - Site Reference ID/Investigator# 29342, Saint Petersburg
  - Site Reference ID/Investigator# 29349, Saint Petersburg
  - Site Reference ID/Investigator# 29457, Saint Petersburg
  - Site Reference ID/Investigator# 29471, Saint Petersburg
  - Site Reference ID/Investigator# 29472, Saint Petersburg
  - Site Reference ID/Investigator# 29473, Saint Petersburg
  - Site Reference ID/Investigator# 29486, Saint Petersburg
  - Site Reference ID/Investigator# 29487, Saint Petersburg
  - Site Reference ID/Investigator# 29488, Saint Petersburg
  - Site Reference ID/Investigator# 29549, Saint Petersburg
  - Site Reference ID/Investigator# 29553, Saint Petersburg
  - Site Reference ID/Investigator# 29554, Saint Petersburg
  - Site Reference ID/Investigator# 29575, Saint Petersburg
  - Site Reference ID/Investigator# 29576, Saint Petersburg
  - Site Reference ID/Investigator# 29584, Saint Petersburg
  - Site Reference ID/Investigator# 29589, Saint Petersburg
  - Site Reference ID/Investigator# 29590, Saint Petersburg
  - Site Reference ID/Investigator# 29592, Saint Petersburg
  - Site Reference ID/Investigator# 29594, Saint Petersburg
  - Site Reference ID/Investigator# 29595, Saint Petersburg
  - Site Reference ID/Investigator# 29611, Saint Petersburg
  - Site Reference ID/Investigator# 29614, Saint Petersburg
  - Site Reference ID/Investigator# 29615, Saint Petersburg
  - Site Reference ID/Investigator# 33322, Saint Petersburg
  - Site Reference ID/Investigator# 6368, Saint Petersburg
  - Site Reference ID/Investigator# 28604, Samara
  - Site Reference ID/Investigator# 28987, Samara
  - Site Reference ID/Investigator# 29183, Samara
  - Site Reference ID/Investigator# 29187, Samara
  - Site Reference ID/Investigator# 29201, Samara
  - Site Reference ID/Investigator# 29202, Samara
  - Site Reference ID/Investigator# 29203, Samara
  - Site Reference ID/Investigator# 29222, Samara
  - Site Reference ID/Investigator# 29253, Samara
  - Site Reference ID/Investigator# 29276, Samara
  - Site Reference ID/Investigator# 29277, Samara
  - Site Reference ID/Investigator# 29474, Samara
  - Site Reference ID/Investigator# 29475, Samara
  - Site Reference ID/Investigator# 29476, Samara
  - Site Reference ID/Investigator# 29523, Samara
  - Site Reference ID/Investigator# 29524, Samara
  - Site Reference ID/Investigator# 29539, Samara
  - Site Reference ID/Investigator# 29540, Samara
  - Site Reference ID/Investigator# 29541, Samara
  - Site Reference ID/Investigator# 29543, Samara
  - Site Reference ID/Investigator# 29616, Samara
  - Site Reference ID/Investigator# 29617, Samara
  - Site Reference ID/Investigator# 29641, Samara
  - Site Reference ID/Investigator# 29643, Samara
  - Site Reference ID/Investigator# 29644, Samara
  - Site Reference ID/Investigator# 29544, Shchëlkovo
  - Site Reference ID/Investigator# 28599, Stavropol
  - Site Reference ID/Investigator# 29005, Stavropol
  - Site Reference ID/Investigator# 29242, Stavropol
  - Site Reference ID/Investigator# 29347, Stavropol
  - Site Reference ID/Investigator# 29348, Stavropol
  - Site Reference ID/Investigator# 29654, Stavropol
  - Site Reference ID/Investigator# 28975, Tolyatti
  - Site Reference ID/Investigator# 29463, Tolyatti
  - Site Reference ID/Investigator# 29572, Tolyatti
  - Site Reference ID/Investigator# 29632, Tolyatti
  - Site Reference ID/Investigator# 29633, Tolyatti
  - Site Reference ID/Investigator# 29094, Tyumen
  - Site Reference ID/Investigator# 29464, Tyumen
  - Site Reference ID/Investigator# 29466, Tyumen
  - Site Reference ID/Investigator# 29656, Tyumen
  - Site Reference ID/Investigator# 29657, Tyumen
  - Site Reference ID/Investigator# 29659, Tyumen
  - Site Reference ID/Investigator# 29661, Tyumen
  - Site Reference ID/Investigator# 29665, Tyumen
  - Site Reference ID/Investigator# 29672, Tyumen
  - Site Reference ID/Investigator# 29677, Tyumen
  - Site Reference ID/Investigator# 33324, Tyumen
  - Site Reference ID/Investigator# 28978, Volgograd
  - Site Reference ID/Investigator# 29250, Volgograd
  - Site Reference ID/Investigator# 29605, Volgograd
  - Site Reference ID/Investigator# 29606, Volgograd
  - Site Reference ID/Investigator# 29607, Volgograd
  - Site Reference ID/Investigator# 29251, Voronezh
  - Site Reference ID/Investigator# 29519, Voronezh
  - Site Reference ID/Investigator# 29521, Voronezh
  - Site Reference ID/Investigator# 29522, Voronezh
  - Site Reference ID/Investigator# 29404, Yekaterinburg
  - Site Reference ID/Investigator# 29405, Yekaterinburg
  - Site Reference ID/Investigator# 29406, Yekaterinburg
  - Site Reference ID/Investigator# 29411, Yekaterinburg
  - Site Reference ID/Investigator# 29412, Yekaterinburg
  - Site Reference ID/Investigator# 29414, Yekaterinburg
- Slovakia (167):
  - Site Reference ID/Investigator# 28754, Banská Bystrica
  - Site Reference ID/Investigator# 28896, Banská Bystrica
  - Site Reference ID/Investigator# 29366, Banská Bystrica
  - Site Reference ID/Investigator# 29367, Banská Bystrica
  - Site Reference ID/Investigator# 28808, Banská Bystrica
  - Site Reference ID/Investigator# 28918, Bardejov
  - Site Reference ID/Investigator# 29129, Bardejov
  - Site Reference ID/Investigator# 29324, Bardejov
  - Site Reference ID/Investigator# 29350, Bardejov
  - Site Reference ID/Investigator# 28932, Bratislava
  - Site Reference ID/Investigator# 28693, Bratislava
  - Site Reference ID/Investigator# 29415, Bratislava
  - Site Reference ID/Investigator# 29417, Bratislava
  - Site Reference ID/Investigator# 28717, Bratislava
  - Site Reference ID/Investigator# 28749, Bratislava
  - Site Reference ID/Investigator# 28614, Bratislava
  - Site Reference ID/Investigator# 29416, Bratislava
  - Site Reference ID/Investigator# 40734, Bratislava
  - Site Reference ID/Investigator# 28849, Bratislava
  - Site Reference ID/Investigator# 28889, Bratislava
  - Site Reference ID/Investigator# 28694, Bratislava
  - Site Reference ID/Investigator# 28745, Bratislava
  - Site Reference ID/Investigator# 28757, Bratislava
  - Site Reference ID/Investigator# 28879, Čierne
  - Site Reference ID/Investigator# 29388, Detva
  - Site Reference ID/Investigator# 29389, Detva
  - Site Reference ID/Investigator# 29357, Dudince
  - Site Reference ID/Investigator# 29358, Dudince
  - Site Reference ID/Investigator# 28880, Dunajská Streda
  - Site Reference ID/Investigator# 29364, Dunajská Streda
  - Site Reference ID/Investigator# 29365, Dunajská Streda
  - Site Reference ID/Investigator# 29312, Galanta
  - Site Reference ID/Investigator# 29313, Galanta
  - Site Reference ID/Investigator# 29380, Galanta
  - Site Reference ID/Investigator# 29381, Galanta
  - Site Reference ID/Investigator# 29056, Hlohovec
  - Site Reference ID/Investigator# 33325, Hlohovec
  - Site Reference ID/Investigator# 29386, Hnúšťa
  - Site Reference ID/Investigator# 29387, Hnúšťa
  - Site Reference ID/Investigator# 28923, Humenné
  - Site Reference ID/Investigator# 29159, Humenné
  - Site Reference ID/Investigator# 29370, Kežmarok
  - Site Reference ID/Investigator# 29371, Kežmarok
  - Site Reference ID/Investigator# 29355, Kežmarok
  - Site Reference ID/Investigator# 29356, Kežmarok
  - Site Reference ID/Investigator# 28907, Kežmarok
  - Site Reference ID/Investigator# 28793, Kolárovo
  - Site Reference ID/Investigator# 29016, Komárno
  - Site Reference ID/Investigator# 28620, Košice
  - Site Reference ID/Investigator# 28621, Košice
  - Site Reference ID/Investigator# 28718, Košice
  - Site Reference ID/Investigator# 28841, Košice
  - Site Reference ID/Investigator# 28909, Košice
  - Site Reference ID/Investigator# 29160, Košice
  - Site Reference ID/Investigator# 29286, Košice
  - Site Reference ID/Investigator# 29287, Košice
  - Site Reference ID/Investigator# 29316, Košice
  - Site Reference ID/Investigator# 29317, Košice
  - Site Reference ID/Investigator# 28762, Košice
  - Site Reference ID/Investigator# 29037, Košice
  - Site Reference ID/Investigator# 28917, Kráľovský Chlmec
  - Site Reference ID/Investigator# 29310, Levice
  - Site Reference ID/Investigator# 29311, Levice
  - Site Reference ID/Investigator# 29292, Levice
  - Site Reference ID/Investigator# 29293, Levice
  - Site Reference ID/Investigator# 28671, Liptovský Hrádok
  - Site Reference ID/Investigator# 29382, Martin
  - Site Reference ID/Investigator# 29383, Martin
  - Site Reference ID/Investigator# 29130, Medzilaborce
  - Site Reference ID/Investigator# 28828, Michalovce
  - Site Reference ID/Investigator# 29284, Modra
  - Site Reference ID/Investigator# 29285, Modra
  - Site Reference ID/Investigator# 28622, Moldava nad Bodvou
  - Site Reference ID/Investigator# 29028, Nitra
  - Site Reference ID/Investigator# 28835, Nitra
  - Site Reference ID/Investigator# 29302, Nitra
  - Site Reference ID/Investigator# 29351, Nová Dubnica
  - Site Reference ID/Investigator# 29352, Nová Dubnica
  - Site Reference ID/Investigator# 29294, Nove Zamke
  - Site Reference ID/Investigator# 29295, Nove Zamke
  - Site Reference ID/Investigator# 29363, Nove Zamke
  - Site Reference ID/Investigator# 29398, Nové Mesto nad Váhom
  - Site Reference ID/Investigator# 29399, Nové Mesto nad Váhom
  - Site Reference ID/Investigator# 29304, Nové Zámky
  - Site Reference ID/Investigator# 29305, Nové Zámky
  - Site Reference ID/Investigator# 29362, Nové Zámky
  - Site Reference ID/Investigator# 28695, Nový Smokovec
  - Site Reference ID/Investigator# 28743, Partizánske
  - Site Reference ID/Investigator# 28744, Pezinok
  - Site Reference ID/Investigator# 28734, Piešťany
  - Site Reference ID/Investigator# 29378, Poprad
  - Site Reference ID/Investigator# 29379, Poprad
  - Site Reference ID/Investigator# 28637, Prešov
  - Site Reference ID/Investigator# 29353, Prešov
  - Site Reference ID/Investigator# 29354, Prešov
  - Site Reference ID/Investigator# 29397, Prešov
  - Site Reference ID/Investigator# 28881, Prievidza
  - Site Reference ID/Investigator# 29314, Prievidza
  - Site Reference ID/Investigator# 29315, Prievidza
  - Site Reference ID/Investigator# 29374, Prievidza
  - Site Reference ID/Investigator# 29375, Prievidza
  - Site Reference ID/Investigator# 29320, Rimavská Sobota
  - Site Reference ID/Investigator# 29321, Rimavská Sobota
  - Site Reference ID/Investigator# 28838, Rožňava
  - Site Reference ID/Investigator# 28761, Ružomberok
  - Site Reference ID/Investigator# 29306, Ružomberok
  - Site Reference ID/Investigator# 29307, Ružomberok
  - Site Reference ID/Investigator# 29372, Ružomberok
  - Site Reference ID/Investigator# 29373, Ružomberok
  - Site Reference ID/Investigator# 28832, Senec
  - Site Reference ID/Investigator# 28897, Senec
  - Site Reference ID/Investigator# 28812, Senica
  - Site Reference ID/Investigator# 28691, Sirk
  - Site Reference ID/Investigator# 28920, Snina
  - Site Reference ID/Investigator# 29083, Snina
  - Site Reference ID/Investigator# 6367, Snina
  - Site Reference ID/Investigator# 28629, Sobrance
  - Site Reference ID/Investigator# 29394, Spišská Nová Ves
  - Site Reference ID/Investigator# 29395, Spišská Nová Ves
  - Site Reference ID/Investigator# 29296, Stará Ľubovňa
  - Site Reference ID/Investigator# 29297, Stará Ľubovňa
  - Site Reference ID/Investigator# 28771, Stará Turá
  - Site Reference ID/Investigator# 29298, Svidník
  - Site Reference ID/Investigator# 29299, Svidník
  - Site Reference ID/Investigator# 28763, Svit
  - Site Reference ID/Investigator# 29308, Šahy
  - Site Reference ID/Investigator# 29309, Šahy
  - Site Reference ID/Investigator# 28638, Šaľa
  - Site Reference ID/Investigator# 28903, Topoľčany
  - Site Reference ID/Investigator# 29282, Topoľčany
  - Site Reference ID/Investigator# 29283, Topoľčany
  - Site Reference ID/Investigator# 29391, Tornaľa
  - Site Reference ID/Investigator# 28919, Trebišov
  - Site Reference ID/Investigator# 28764, Trenčianske Teplice
  - Site Reference ID/Investigator# 29119, Trenčín
  - Site Reference ID/Investigator# 28806, Trenčín
  - Site Reference ID/Investigator# 29133, Trenčín
  - Site Reference ID/Investigator# 28667, Trnava
  - Site Reference ID/Investigator# 28805, Trnava
  - Site Reference ID/Investigator# 28892, Trnava
  - Site Reference ID/Investigator# 28910, Trnava
  - Site Reference ID/Investigator# 28929, Trnava
  - Site Reference ID/Investigator# 29359, Trnava
  - Site Reference ID/Investigator# 29360, Trnava
  - Site Reference ID/Investigator# 29384, Trnava
  - Site Reference ID/Investigator# 29385, Trnava
  - Site Reference ID/Investigator# 29288, Turčianske Teplice
  - Site Reference ID/Investigator# 29289, Turčianske Teplice
  - Site Reference ID/Investigator# 28690, Turzovka
  - Site Reference ID/Investigator# 28716, Veľké Kapušany
  - Site Reference ID/Investigator# 28921, Veľké Zálužie
  - Site Reference ID/Investigator# 28819, Veľký Biel
  - Site Reference ID/Investigator# 28883, Veľký Krtíš
  - Site Reference ID/Investigator# 29368, Vranov nad Topľou
  - Site Reference ID/Investigator# 29369, Vranov nad Topľou
  - Site Reference ID/Investigator# 29303, Vráble
  - Site Reference ID/Investigator# 29023, Vrútky
  - Site Reference ID/Investigator# 28688, Zavar
  - Site Reference ID/Investigator# 29318, Zlaté Moravce
  - Site Reference ID/Investigator# 29319, Zlaté Moravce
  - Site Reference ID/Investigator# 28736, Žiar nad Hronom
  - Site Reference ID/Investigator# 28686, Žilina
  - Site Reference ID/Investigator# 28829, Žilina
  - Site Reference ID/Investigator# 29290, Žilina
  - Site Reference ID/Investigator# 29291, Žilina
  - Site Reference ID/Investigator# 29322, Žilina
  - Site Reference ID/Investigator# 29323, Žilina
- Slovenia (130):
  - Site Reference ID/Investigator# 30484, Adjovscina
  - Site Reference ID/Investigator# 30485, Adjovscina
  - Site Reference ID/Investigator# 6366, Adjovscina
  - Site Reference ID/Investigator# 33326, Bled
  - Site Reference ID/Investigator# 33327, Bled
  - Site Reference ID/Investigator# 28625, Celje
  - Site Reference ID/Investigator# 29033, Celje
  - Site Reference ID/Investigator# 29837, Celje
  - Site Reference ID/Investigator# 30486, Celje
  - Site Reference ID/Investigator# 30487, Celje
  - Site Reference ID/Investigator# 28587, Cerknica
  - Site Reference ID/Investigator# 33328, Cerknica
  - Site Reference ID/Investigator# 30088, Deskle
  - Site Reference ID/Investigator# 30145, Dol pri Hrastniku
  - Site Reference ID/Investigator#28729, Dolenjske Toplice
  - Site Reference ID/Investigator# 28775, Domžale
  - Site Reference ID/Investigator# 30186, Fram
  - Site Reference ID/Investigator# 29918, Golnik
  - Site Reference ID/Investigator# 33331, Golnik
  - Site Reference ID/Investigator# 29040, Grosuplje
  - Site Reference ID/Investigator# 30488, Grosuplje
  - Site Reference ID/Investigator# 29955, Ilirska Bistrica
  - Site Reference ID/Investigator# 30490, Jesenice
  - Site Reference ID/Investigator# 30491, Jesenice
  - Site Reference ID/Investigator# 30492, Jesenice
  - Site Reference ID/Investigator# 28689, Koper
  - Site Reference ID/Investigator# 30164, Kostanjevica na Krki
  - Site Reference ID/Investigator# 29438, Kranj
  - Site Reference ID/Investigator# 29439, Kranj
  - Site Reference ID/Investigator# 30204, Kranj
  - Site Reference ID/Investigator# 30494, Kranj
  - Site Reference ID/Investigator# 30495, Kranj
  - Site Reference ID/Investigator# 30496, Kranj
  - Site Reference ID/Investigator# 30000, Kropa
  - Site Reference ID/Investigator# 29168, Krško
  - Site Reference ID/Investigator# 29821, Krško
  - Site Reference ID/Investigator# 30117, Limbuš
  - Site Reference ID/Investigator# 28720, Litija
  - Site Reference ID/Investigator# 28884, Litija
  - Site Reference ID/Investigator# 28727, Ljubljana
  - Site Reference ID/Investigator# 28779, Ljubljana
  - Site Reference ID/Investigator# 29015, Ljubljana
  - Site Reference ID/Investigator# 29171, Ljubljana
  - Site Reference ID/Investigator# 29751, Ljubljana
  - Site Reference ID/Investigator# 29996, Ljubljana
  - Site Reference ID/Investigator# 30012, Ljubljana
  - Site Reference ID/Investigator# 30199, Ljubljana
  - Site Reference ID/Investigator# 30498, Ljubljana
  - Site Reference ID/Investigator# 30499, Ljubljana
  - Site Reference ID/Investigator# 30500, Ljubljana
  - Site Reference ID/Investigator# 30501, Ljubljana
  - Site Reference ID/Investigator# 30502, Ljubljana
  - Site Reference ID/Investigator# 30503, Ljubljana
  - Site Reference ID/Investigator# 28715, Ljutomer
  - Site Reference ID/Investigator# 30120, Ljutomer
  - Site Reference ID/Investigator# 30505, Logatec
  - Site Reference ID/Investigator# 28930, Maribor
  - Site Reference ID/Investigator# 29460, Maribor
  - Site Reference ID/Investigator# 29461, Maribor
  - Site Reference ID/Investigator# 29679, Maribor
  - Site Reference ID/Investigator# 30017, Maribor
  - Site Reference ID/Investigator# 30018, Maribor
  - Site Reference ID/Investigator# 30128, Maribor
  - Site Reference ID/Investigator# 30221, Maribor
  - Site Reference ID/Investigator# 30507, Maribor
  - Site Reference ID/Investigator# 30508, Maribor
  - Site Reference ID/Investigator# 28640, Markovci
  - Site Reference ID/Investigator# 2392, Mežica
  - Site Reference ID/Investigator# 28642, Miklavž na Dravskem Polju
  - Site Reference ID/Investigator# 28951, Murska Sobota
  - Site Reference ID/Investigator# 30005, Murska Sobota
  - Site Reference ID/Investigator# 30081, Murska Sobota
  - Site Reference ID/Investigator# 30196, Muta
  - Site Reference ID/Investigator# 28952, Naklo
  - Site Reference ID/Investigator# 30087, Nazarje
  - Site Reference ID/Investigator# 28958, Nova Gorica
  - Site Reference ID/Investigator# 28959, Novo Mesto
  - Site Reference ID/Investigator# 30142, Novo Mesto
  - Site Reference ID/Investigator# 30125, Oplotnica
  - Site Reference ID/Investigator# 30509, Ormož
  - Site Reference ID/Investigator# 30510, Ormož
  - Site Reference ID/Investigator# 30131, Polzela
  - Site Reference ID/Investigator# 29920, Postojna
  - Site Reference ID/Investigator# 30119, Postojna
  - Site Reference ID/Investigator# 30511, Prevalje
  - Site Reference ID/Investigator# 30512, Prevalje
  - Site Reference ID/Investigator# 28810, Ptuj
  - Site Reference ID/Investigator# 28850, Ptuj
  - Site Reference ID/Investigator# 28983, Ptuj
  - Site Reference ID/Investigator# 30147, Ptuj
  - Site Reference ID/Investigator# 30123, Puconci
  - Site Reference ID/Investigator# 33329, Radeče
  - Site Reference ID/Investigator# 29906, Radenci
  - Site Reference ID/Investigator# 28985, Radovljica
  - Site Reference ID/Investigator# 30124, Radovljica
  - Site Reference ID/Investigator# 30095, Ravne na Koroškem
  - Site Reference ID/Investigator# 30513, Ravne na Koroškem
  - Site Reference ID/Investigator# 30514, Ravne na Koroškem
  - Site Reference ID/Investigator# 30135, Ribnica
  - Site Reference ID/Investigator# 33330, Rogaška Slatina
  - Site Reference ID/Investigator# 28885, Ruše
  - Site Reference ID/Investigator# 30162, Senovo
  - Site Reference ID/Investigator# 30015, Sevnica
  - Site Reference ID/Investigator# 30113, Sevnica
  - Site Reference ID/Investigator# 30168, Sevnica
  - Site Reference ID/Investigator# 30517, Sevnica
  - Site Reference ID/Investigator# 30518, Sevnica
  - Site Reference ID/Investigator# 30130, Sežana
  - Site Reference ID/Investigator# 29125, Sladki Vrh
  - Site Reference ID/Investigator# 28825, Slovenska Bistrica
  - Site Reference ID/Investigator# 28994, Slovenske Konjice
  - Site Reference ID/Investigator# 28641, Straža
  - Site Reference ID/Investigator# 28738, Šentilj v Slovenskih goricah
  - Site Reference ID/Investigator# 28609, Šentjur pri Celju
  - Site Reference ID/Investigator# 30163, Šentjur pri Celju
  - Site Reference ID/Investigator# 28851, Škofljica
  - Site Reference ID/Investigator# 29917, Šoštanj
  - Site Reference ID/Investigator# 29090, Tolmin
  - Site Reference ID/Investigator# 30519, Trebnje
  - Site Reference ID/Investigator# 30520, Trebnje
  - Site Reference ID/Investigator# 29093, Turnišče
  - Site Reference ID/Investigator# 29098, Velenje
  - Site Reference ID/Investigator# 29045, Vojnik
  - Site Reference ID/Investigator# 30121, Vrhnika
  - Site Reference ID/Investigator# 28618, Zagorje
  - Site Reference ID/Investigator# 30144, Zagorje
  - Site Reference ID/Investigator# 29106, Zreče
  - Site Reference ID/Investigator# 30195, Zreče
  - Site Reference ID/Investigator# 28639, Žalec
  - Site Reference ID/Investigator# 30187, Žalec
- Ukraine (50):
  - Site Reference ID/Investigator# 10476, Dnipropetrovsk
  - Site Reference ID/Investigator# 30523, Dnipropetrovsk
  - Site Reference ID/Investigator# 30524, Dnipropetrovsk
  - Site Reference ID/Investigator# 30525, Dnipropetrovsk
  - Site Reference ID/Investigator# 30526, Dnipropetrovsk
  - Site Reference ID/Investigator# 30527, Donetsk
  - Site Reference ID/Investigator# 30528, Donetsk
  - Site Reference ID/Investigator# 30529, Donetsk
  - Site Reference ID/Investigator# 30530, Donetsk
  - Site Reference ID/Investigator# 30541, Kharkiv
  - Site Reference ID/Investigator# 30542, Kharkiv
  - Site Reference ID/Investigator# 30543, Kharkiv
  - Site Reference ID/Investigator# 30544, Kharkiv
  - Site Reference ID/Investigator# 30636, Kiev
  - Site Reference ID/Investigator# 30637, Kiev
  - Site Reference ID/Investigator# 30638, Kiev
  - Site Reference ID/Investigator# 30639, Kiev
  - Site Reference ID/Investigator# 30640, Kiev
  - Site Reference ID/Investigator# 30641, Kiev
  - Site Reference ID/Investigator# 30642, Kiev
  - Site Reference ID/Investigator# 30643, Kiev
  - Site Reference ID/Investigator# 30644, Kiev
  - Site Reference ID/Investigator# 30645, Kiev
  - Site Reference ID/Investigator# 30646, Kiev
  - Site Reference ID/Investigator# 30647, Kiev
  - Site Reference ID/Investigator# 30546, Luhansk
  - Site Reference ID/Investigator# 30547, Luhansk
  - Site Reference ID/Investigator# 30548, Luhansk
  - Site Reference ID/Investigator# 30545, Luhansk
  - Site Reference ID/Investigator# 30549, Lviv
  - Site Reference ID/Investigator# 30550, Lviv
  - Site Reference ID/Investigator# 30551, Lviv
  - Site Reference ID/Investigator# 30552, Lviv
  - Site Reference ID/Investigator# 30610, Odesa
  - Site Reference ID/Investigator# 30611, Odesa
  - Site Reference ID/Investigator# 30612, Odesa
  - Site Reference ID/Investigator# 30613, Odesa
  - Site Reference ID/Investigator# 30634, Sevastopol
  - Site Reference ID/Investigator# 30635, Sevastopol
  - Site Reference ID/Investigator# 30607, Simferopol
  - Site Reference ID/Investigator# 30608, Simferopol
  - Site Reference ID/Investigator# 30609, Simferopol
  - Site Reference ID/Investigator# 30648, Vinnitsa
  - Site Reference ID/Investigator# 30649, Vinnitsa
  - Site Reference ID/Investigator# 30650, Vinnitsa
  - Site Reference ID/Investigator# 30651, Vinnitsa
  - Site Reference ID/Investigator# 30596, Zaporizhzhya
  - Site Reference ID/Investigator# 30597, Zaporizhzhya
  - Site Reference ID/Investigator# 30598, Zaporizhzhya
  - Site Reference ID/Investigator# 30599, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15,873 participants enrolled in the study. Of these, documentation was available for 15,436 participants. 743 participants were excluded for the following reasons: No Tarka therapy documentation (739) and no follow-up data provided (4), leaving a study population of 14,693. No group assignments were made as the study design was observational.
Groups:
- Tarka Therapy: Tarka (trandolapril/verapamil hydrochloride) was to be prescribed in a routine manner according to the terms of local regulatory authorizations. Eligible participants had a high risk of developing diabetes mellitus and high blood pressure that was not controlled with a single medication. Participants were to be treated by secondary care specialists such as internal medicine specialists, nephrologists, and endocrinologists.
Period: Overall Study
Arm/Group | Tarka Therapy
Started | 15873
Completed | 14442
Not Completed | 1431
Not completed — No Documentation of Tarka Therapy | 739
Not completed — No Documentation Available | 437
Not completed — Adverse Event | 157
Not completed — Reason Unknown | 39
Not completed — Withdrawal by Subject | 18
Not completed — Financial Reasons | 15
Not completed — Lack of Effectiveness | 12
Not completed — Physician Decision | 4
Not completed — Improved Status of Participant | 4
Not completed — No Follow-up Documentation Available | 4
Not completed — Non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tarka Therapy
Number analyzed (Participants) | 14693
Age Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.5)
Age, Customized [Number; unit: participants]
  18 years of age or younger | 2
  Over 18 and less than 65 | 10565
  65 and older | 4085
  Age not reported | 41
Sex/Gender, Customized [Number; unit: participants]
  Female | 7559
  Male | 7034
  Gender not reported | 100
Region of Enrollment [Number; unit: participants]
  Bulgaria | 309
  Czech Republic | 5643
  Romania | 1251
  Russian Federation | 2085
  Slovakia | 3179
  Slovenia | 1238
  Ukraine | 988
Time Since Diagnosis of Essential Hypertension [Number; unit: participants]
  At study inclusion | 249
  Less than 1 year | 108
  Between 1 and 2 years | 1536
  Between 2 and 3 years | 1573
  Between 3 and 5 years | 2482
  Between 5 and 10 years | 4187
  10 years or more | 4153
  Time since diagnosis not reported | 405
Risk Factors for Developing Diabetes [Number; unit: participants]
  Positive Family History of Diabetes | 2891
  Obesity | 3661
  Impaired Fasting Glucose (IFG) | 506
  Positive Family History and Obesity | 2983
  Positive Family History and IFG | 563
  Obesity and IFG | 1344
  Positive Family History, Obesity, and IFG | 1091
  Diabetes | 288
  Risk factors not reported | 1366
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (4.8)
Body Weight [Mean (Standard Deviation); unit: kg] | 87.1 (15.2)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 97.8 (13.1)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Systolic Blood Pressure and Diastolic Blood Pressure From Baseline to Study End
Description: Participants were to be followed for 6 months. Changes in systolic and diastolic blood pressure were assessed by comparing the blood pressure measurements obtained at the end of Tarka treatment (approximately 6 months) to baseline values. For this analysis of effectiveness the last available value was considered the analysis time point "end of study".
Time Frame: Baseline to 6 months/study end
Population: 2122 participants were excluded from this analysis for the following reasons: age less than 18 years (1), no diagnosis of hypertension (18), not at risk for diabetes (1650), no follow-up blood pressure values (48), no baseline blood pressure values (360), and started Tarka at/after first follow-up visit (45).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tarka Therapy
Number analyzed (Participants) | 12571
mmHg
  Systolic blood pressure change from baseline | -28.5 (14.8)
  Diastolic blood pressure change from baseline | -16.1 (9.5)

2. Secondary Outcome: Percentage of Participants Achieving Target Blood Pressure (Less Than 140/90) at Study End and the Need for Other Antihypertensive Drugs, Clustered by Type(s) of Drugs Added to Tarka.
Description: The percentages of participants achieving and not achieving the target blood pressure of less than 140/90 mmHg at the end of the study are presented. Percentages of participants taking Tarka only or taking Tarka plus another antihypertensive drug are summarized by type of drug: beta blockers, angiotensin-converting enzyme (ACE) inhibitors, calcium antagonists, diuretics, and angiotensin II (AT-II) receptor antagonists. Participants taking drugs that did not fit any of the above groups (Other), unknown drugs (Unknown), or more than one additional antihypertensive agent are also summarized.
Time Frame: 6 months
Population: 2122 participants were excluded from the analysis for the following reasons: age less than 18 years (1), no diagnosis of hypertension (18), not at risk for diabetes (1650), no follow-up blood pressure values (48), no baseline blood pressure values (360), and started Tarka at/after first follow-up visit (45).
Measure: Number; unit: Percentage of participants
Arm/Group | Tarka Therapy
Number analyzed (Participants) | 12571
Percentage of participants
  Achieved target blood pressure | 68.1
  Did not achieve target blood pressure | 31.9
  Taking Tarka only | 74.6
  Taking Tarka and 1 antihypertensive drug | 20.5
  Taking Tarka and a beta blocking agent | 1.1
  Taking Tarka and an ACE-inhibitor | 1.4
  Taking Tarka and a calcium antagonist | 0.9
  Taking Tarka and a diuretic | 10.7
  Taking Tarka and an AT-II receptor antagonist | 0.8
  Taking Tarka and 1 Other antihypertensive drug | 4.2
  Taking Tarka and an Unknown antihypertensive drug | 1.3
  Taking Tarka and more than 1 antihypertensive drug | 4.9

3. Secondary Outcome: Evaluation of Adverse Events (AEs) Leading to Discontinuation of Tarka and a Summary of All AEs Possibly or Probably Related to Tarka by Frequency and Severity
Description: The number of AEs leading to Tarka discontinuation are summarized. AEs that were considered by the investigator to be possibly or probably related to Tarka are summarized by the severity of the AE (classified as mild, moderate, or severe). AEs considered possibly or probably related to Tarka that led to the discontinuation of Tarka are also presented by severity.
Time Frame: 6 months
Population: This analysis used the safety analysis population, which included any participant who took at least one dose of Tarka and had at least one follow-up visit.
Measure: Number; unit: Events
Arm/Group | Tarka Therapy
Number analyzed (Participants) | 14693
Events
  Any AE that led to discontinuation (d/c) of Tarka | 224
  AEs possibly or probably related to Tarka | 199
  a) Severity: Mild | 107
  b) Severity: Moderate | 82
  c) Severity: Severe | 5
  d) Severity: Unknown | 5
  Any AE possibly/probably related that led to d/c | 171
  a) Severity: Mild | 85
  b) Severity: Moderate | 79
  c) Severity: Severe | 5
  d) Severity: Unknown | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tarka Therapy
Serious Adverse Events (participants affected / at risk) | 16/14693
Other Adverse Events (participants affected / at risk) | 0/15873
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tarka Therapy (N=14693)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 11 (11)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.